CLINICAL TRIAL: NCT05918185
Title: The Role of the Comprehensive Geriatric Assessment in Elderly Patients With Multiple Myeloma: A Single Center Prospective Study
Brief Title: Evaluation of Comprehensive Geriatric Assessment and Laboratory Biomarkers in Elderly Patients With Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 21-010499; NCI-2022-06872 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-010499 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2023-05-17; First posted 2023-06-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Specimen Handling; Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (Surveys, cGA, blood sample, EHR review): Patients complete surveys and undergo cGA, blood sample collection, and EHR review on study.
  Interventions: Procedure: Biospecimen Collection; Other: Comprehensive Geriatric Assessment; Other: Electronic Health Record Review; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Comprehensive Geriatric Assessment — Undergo cGA
Other: Electronic Health Record Review — Medical records are reviewed
Other: Survey Administration — Complete surveys

SUMMARY:
This study evaluates the association between a comprehensive geriatric assessment and laboratory biomarkers with the side effects of chemotherapy in older patients with multiple myeloma (MM). The comprehensive geriatric assessment is a tool that can help to determine how fit a patient is. It is composed of a series of questions and tests designed for older people to evaluate their physical function, mental status, mental health, nutritional status, social support, level of social activity, and the presence of other medical problems. In addition to geriatric assessment domains, laboratory biomarkers may provide information on physiologic dysfunction as a measure for evaluation of frailty in the cancer setting. This study will help researchers in the future by predicting which patients will have more side effects with chemotherapy based on their comprehensive geriatric assessment and laboratory biomarkers, which will allow adjustments to treatment in older adult patients with MM.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the association between a baseline comprehensive geriatric assessment (cGA) and chemotherapy toxicity in the first 4 months of treatment measured by treatment-related adverse events, patient-reported outcomes (PROs), and treatment discontinuation in older patients (>= 65 years) with multiple myeloma (MM).

SECONDARY OBJECTIVES:

I. To evaluate the association between a baseline cGA and baseline disease- and host- related laboratory characteristics and cytogenetic risk profile by fluorescence in situ hybridization among newly diagnosed older (>= 65 years) patients with MM.

II. To evaluate how the cGA changes over 4 months from the start of treatment and the association between those changes and treatment response in older patients (>= 65 years) with MM.

III. To evaluate the association between proposed frailty biomarkers at baseline and treatment toxicity in the first 4 months of treatment measured by treatment-related adverse events, PROs, and treatment discontinuation in older (>= 65 years) patients with MM.

OUTLINE: This is an observational study.

Patients complete surveys and undergo cGA, blood sample collection, and electronic health record (EHR) review on study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 65 years
* Diagnosis of MM based on International Myeloma Working Group (IMWG) diagnostic criteria
* Newly diagnosed or have received 1 prior line of treatment
* Planned to start a new treatment for MM within 30 days
* Transplant eligible or ineligible
* Fluent in English (all assessment tools are in English)
* Able to provide written informed consent

Exclusion Criteria:

* Received > 1 prior line of treatment
* Patients included in an interventional therapeutic trial
* Not able to give informed consent
* Severe mental or cognitive disorder precluding geriatric assessment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over the age of 65 planned to start a new treatment for MM at Mayo Clinic in Rochester.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | Up to 4 months
  Will graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The maximum observed grade per adverse event and capture grade >= 3 toxicities.

SECONDARY OUTCOMES:
Chemotherapy toxicity | Up to 4 months
  Will be analyzed longitudinally using toxicity over time analysis which measures adverse events over time, providing information on timing and evolution of symptoms during treatment.
Patient reported outcome (PRO) questionnaire | Up to 4 months
  Will be assessed at the end of each treatment cycle (prior to each new cycle) at scheduled visits for a total of 4 months or until treatment discontinuation whichever comes first using the PRO Measurement Information System Global Health which is a 10-item questionnaire that assesses a patient's global heath. All questions have a five-point Likert-type scale, except for the rating of pain question which has a 10-point scale. Subscale scores can be generated for Global Physical Health and Global Mental for each patient.
Patient reported outcome (PRO-CTCAE) questionnaire | Up to 4 months
  Select PRO-CTCAE symptomatic adverse event items to assess the presence, severity and interference of symptoms experienced by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Shaji K. Kumar, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials